CLINICAL TRIAL: NCT00524875
Title: Effect of Intravitreal Bevacizumab on Early Post-Vitrectomy Hemorrhage in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8657
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-08

CONDITIONS: Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; Bevacizumab; Early post-vitrectomy vitreous hemorrhage
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intravitreal bevacizumab injection 1-2 weeks before surgery
  Interventions: Drug: Bevacizumab
- 2 (Sham Comparator): Sham injection (needleless syringe pressed against conjunctiva)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — One dose of bevacizumab (1.25 mg/0.05 cc) one to two weeks before pars plana vitrectomy for diabetic retinopathy

SUMMARY:
The purpose of this study is to determine whether bevacizumab 1-2 weeks before vitrectomy is effective in lowering the rate of early post-vitrectomy vitreous hemorrhage in diabetic patients.

DETAILED DESCRIPTION:
Diabetes is the leading cause of blindness in the age range of 20-64 years. Pars plana vitrectomy may be indicated for the management of advanced proliferative diabetic retinopathy. Early post-vitrectomy hemorrhage in diabetic patients is relatively common; it occurs in 29% -75% of patients in the first month after surgery. This may cause delayed visual rehabilitation and detection of surgical complications such as retinal break or detachment. Preliminary reports such as case series reported by Spaide RF, et al showed beneficial effect of bevacizumab in proliferative diabetic retinopathy complicated by vitreous hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* All eyes who are candidate for pars plana vitrectomy because of complications of diabetic retinopathy such as nonclearing vitreous hemorrhage, tractional retinal detachment threatening macula, active progressive PDR

Exclusion Criteria:

* One eye patient
* Best corrected visual acuity better than 20/50
* Pregnancy
* Use of internal tamponade such as silicone oil during surgery
* Concurrent ophthalmic surgery such as cataract extraction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-01; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
early post-vitrectomy vitreous hemorrhage

SECONDARY OUTCOMES:
Visual improvement

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran